CLINICAL TRIAL: NCT00123734
Title: Phase II Clinical Trial to Evaluate the Accuracy of Anti-Fibrin Humanized Monoclonal Antibody (DI-DD3B6/22-80B3) Fab' Protein Fragment (ThromboView) Conjugated With Technetium-99m in the Detection of Deep Vein Thrombosis
Brief Title: Clinical Trial to Evaluate the Accuracy of [99mTc] ThromboView in the Detection of Deep Vein Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agen Biomedical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAN/US-001-II-DVT
Record Dates: First submitted 2005-07-24; First posted 2005-07-26 (Estimated); Results first posted 2009-08-24 (Estimated); Last update posted 2009-08-24 (Estimated); Status verified 2009-07

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — thromboview

INTERVENTIONS:
Drug: ThromboView

SUMMARY:
The assessment of patients with suspected deep vein thrombosis (DVT) is a common clinical scenario that, despite major advances in diagnostic testing, continues to be challenging.

The diagnosis of DVT remains problematic in:

* patients with suspected first DVT who have a moderate or high pre-test probability (PTP) for DVT and a normal compression ultrasound (CUS);
* patients with suspected recurrent DVT; and
* patients in whom CUS or contrast venography is technically difficult or not feasible due to patient characteristics.

In patients with suspected first DVT who have a moderate or high PTP and a normal CUS, DVT occurs in up to 10% of cases. Thus, additional diagnostic testing is required, such as venography or serial CUS, so that DVT is not missed, but these approaches are costly and invasive.

In patients with suspected recurrent DVT, currently used diagnostic approaches are problematic because they all have limitations in differentiating old disease from true recurrent disease.

CUS is technically difficult in selected patients, particularly those who are obese.

Contrast venography is the gold standard diagnostic test for DVT to which all other diagnostic venous imaging modalities for DVT are compared and judged. The Food and Drug Administration (FDA) requires that a new diagnostic test for DVT be assessed against venography.

[99mTc] ThromboView® is a novel diagnostic test based on a 99mTc-labeled monoclonal antibody specific for D-dimer fragments of cross-linked fibrin that are found in acute DVT. After intravenous injection of [99mTc] ThromboView®, there is uptake of the monoclonal antibody by acute, D-dimer rich, venous thrombi. This is visualized with nuclear medicine imaging as an area of increased radioisotope activity that corresponds to the location of DVT.

Based on the biologic and imaging characteristics of [99mTc] ThromboView®, this diagnostic test has the potential to:

* identify small non-occlusive proximal DVT or distal DVT in patients with a moderate or high PTP and normal CUS;
* differentiate old from new DVT in patients with suspected recurrent DVT;
* diagnose or exclude DVT in patients in whom CUS is not technically feasible; and
* provide an alternative to venography that is non-invasive, has no contrast-related toxicity and is easily administered.

The present study is the first phase II clinical trial of [99mTc] ThromboView® in patients with suspected initial or recurrent DVT in whom DVT has been confirmed or excluded by venography. A phase II clinical trial to investigate the diagnostic accuracy of [99mTc] ThromboView® is justified because:

* ThromboView® was well tolerated, with no significant toxicity in studies involving animals and healthy volunteers; and
* it has shown promise in Phase I trials as a non-invasive diagnostic test for acute DVT.

ELIGIBILITY:
Inclusion Criteria:

* Adult man or woman, aged ≥18 years, presenting with suspected lower-limb initial or recurrent DVT.
* Moderate or high pre-test probability (PTP) for DVT.
* Onset of symptoms occurred within the last 7 days.
* Women of childbearing potential to have a negative pregnancy test as determined by measuring serum β-hCG levels at time of study enrolment.

Exclusion Criteria:

* Receiving anticoagulant therapy at therapeutic doses for >3 days.
* Life expectancy <3 months.
* Patient with a renal transplant.
* Renal dysfunction: serum creatinine >1.5x upper limit of normal range.
* Hepatic dysfunction: serum transaminases >3x upper limit of normal range.
* Current pregnancy or lactation; or conception intended within 90 days of enrolment
* Of childbearing potential and unwilling to use adequate contraception for 30 days following enrolment
* Unable to undergo lower limb ascending venography on symptomatic leg(s).
* Allergy or other contraindication to intravenous contrast dye.
* Prior exposure to murine or humanized antibodies.
* Prior imaging studies with: I131 within the last month; In111 or Ga67 within the last 2 weeks; Tc99m labelled RBCs, WBCs or albumin within the last 48 hours; Tc99m or F18 within the last 24 hours; prior non-imaging, non-therapeutic nuclear medicine studies with I131 (eg., 24-hour RAI uptake) within the last 2 weeks.
* Previous participation in the present study.
* Geographic inaccessibility that precludes follow-up visits.
* Patient is unwilling or unable to provide informed consent.
* Patient is unsuitable for the study, at the Study Investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-03; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Jim Douketis, MD FRCPC, Principal Investigator — Hamilton Health Sciences Corporation; Jeff Ginsberg, MD FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (12):
- United States (5):
  - UC Davis, Sacramento, California
  - UCSD Medical Centre, San Diego, California
  - Henry Ford Hospital, Detroit, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma, Health Sciences Center, Oklahoma City, Oklahoma
- Canada (7):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University, Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Henderson General Site, Hamilton, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hotel-Dieu Du CHUM, Montreal, Quebec
  - Centre hospitalier de L'Universite Laval, Sainte-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 94 participants were enrolled into the study. The first participant was enrolled on 4 March 2005, and the last participant was enrolled on 6 February 2006. All participants were enrolled in hosptial.
Pre-assignment Details: 12 participants did not recieve study drug (6 had no venography, 3 withdrew consent, 2 had an alternate diagnosis and 1 was a dropout).
Period: Overall Study
Arm/Group | Group 1
Started | 82
Completed | 74
Not Completed | 8
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — Dropout | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 55.12 (15.148)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: To Provide Estimates of the Specificity of [99mTc] ThromboView® in Patients With Excluded Initial DVT
Time Frame: May 2007
Population: Number of participants with suspected initial DVT with evaluable images
Measure: Mean (95% Confidence Interval); unit: % Specificity
Groups:
- 1 Hour Image Set: Review of whole leg 1 hour images
- 3 Hour Image Set: Review of 3 hour whole leg images
- 15 Min and 1 Hour Image Set: Review of whole leg 15 minute and 1 hour images in combination
- 15 Minute and 3 Hour Image Set: Review of whole leg 15 minute and 3 hour images in combination
Arm/Group | 1 Hour Image Set | 3 Hour Image Set | 15 Min and 1 Hour Image Set | 15 Minute and 3 Hour Image Set
Number analyzed (Participants) | 26 | 26 | 26 | 26
% Specificity | 76.9 [58.0 to 89.0] | 65.4 [46.2 to 80.6] | 100 [87.1 to 100] | 96.2 [81.1 to 99.3]

2. Secondary Outcome: To Provide Estimates of the Specificity of [99mTc] ThromboView® in Patients With Suspected Recurrent DVT in Whom Disease Recurrence Has Been Excluded
Time Frame: May 2007
Population: Number of participants with suspected recurrent DVT with evaluable images
Measure: Mean (95% Confidence Interval); unit: % Specificity
Arm/Group | 1 Hour Image Set | 3 Hour Image Set | 15 Min and 1 Hour Image Set | 15 Minute and 3 Hour Image Set
Number analyzed (Participants) | 11 | 11 | 11 | 11
% Specificity | 36.4 [15.2 to 64.6] | 72.7 [43.4 to 90.3] | 63.6 [35.4 to 84.8] | 72.7 [43.4 to 90.3]

3. Secondary Outcome: To Provide Estimates of the Specificity of [99mTc] ThromboView® for Imaging Suspected Proximal Initial DVT
Time Frame: May 2007
Population: Number of participants with suspected initial DVT with evaluable images
Measure: Mean (95% Confidence Interval); unit: % Specificity
Arm/Group | 1 Hour Image Set | 3 Hour Image Set | 15 Min and 1 Hour Image Set | 15 Minute and 3 Hour Image Set
Number analyzed (Participants) | 29 | 30 | 29 | 30
% Specificity | 86.2 [69.4 to 94.5] | 70.0 [52.1 to 83.3] | 100 [88.3 to 100] | 96.7 [83.3 to 99.4]

4. Secondary Outcome: To Provide Estimates of the Sensitivity of [99mTc] ThromboView® for Imaging Suspected Proximal Initial DVT
Time Frame: May 2007
Population: Number of participants with suspected initial DVT with evaluable images
Measure: Mean (95% Confidence Interval); unit: % Sensitivity
Arm/Group | 1 Hour Image Set | 3 Hour Image Set | 15 Min and 1 Hour Image Set | 15 Minute and 3 Hour Image Set
Number analyzed (Participants) | 19 | 20 | 19 | 19
% Sensitivity | 42.1 [23.1 to 63.7] | 90.0 [69.9 to 97.2] | 15.8 [5.5 to 37.6] | 84.2 [62.4 to 94.5]

5. Primary Outcome: To Provide Estimates of the Sensitivity of [99mTc] ThromboView® in Patients With Confirmed Initial DVT.
Time Frame: September 2005
Measure: Mean (95% Confidence Interval); unit: % Sensitivity
Arm/Group | 1 Hour Image Set | 3 Hour Image Set | 15 Min and 1 Hour Image Set | 15 Minute and 3 Hour Image Set
Number analyzed (Participants) | 27 | 27 | 27 | 27
% Sensitivity | 37.0 [21.5 to 55.8] | 74.1 [55.3 to 86.8] | 11.1 [3.9 to 28.1] | 59.3 [40.7 to 75.5]

6. Secondary Outcome: To Provide Estimates of the Specificity of [99mTc] ThromboView® for Imaging Suspected Distal Initial DVT
Time Frame: May 2007
Population: Number of participants with suspected initial DVT with evaluable images
Measure: Mean (95% Confidence Interval); unit: % Specificity
Arm/Group | 1 Hour Image Set | 3 Hour Image Set | 15 Min and 1 Hour Image Set | 15 Minute and 3 Hour Image Set
Number analyzed (Participants) | 29 | 29 | 29 | 29
% Specificity | 93.1 [78.0 to 98.1] | 89.7 [73.6 to 96.4] | 100 [88.3 to 100] | 96.6 [82.8 to 99.4]

7. Secondary Outcome: To Provide Estimates of the Sensitivity of [99mTc] ThromboView® for Imaging Suspected Distal Initial DVT
Time Frame: May 2007
Population: Number of participants with suspected initial DVT with evaluable images
Measure: Mean (95% Confidence Interval); unit: % Sensitivity
Arm/Group | 1 Hour Image Set | 3 Hour Image Set | 15 Min and 1 Hour Image Set | 15 Minute and 3 Hour Image Set
Number analyzed (Participants) | 22 | 22 | 22 | 22
% Sensitivity | 18.2 [7.3 to 38.5] | 40.9 [23.3 to 61.3] | 0 [0.0 to 14.9] | 36.4 [19.7 to 57.1]

8. Secondary Outcome: To Provide Estimates of the Sensitivity and Specificity of [99mTc] ThromboView® for DVT at the 1-hour and 3-hour Imaging Time Points
Time Frame: May 2007
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days